CLINICAL TRIAL: NCT05347355
Title: Comparison of Spencer Technique and Gongs Mobilization on Pain, Range of Motion, Disability and Scapular Symmetry in Patients With Phase ii Adhesive Capsulitis
Brief Title: Comparison of Spencer Technique and Gongs Mobilization in Patients With Phase ii Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0130 Nimra
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive; scapula; mobilization; glenohumeral joint
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spencer technique along with conventional treatment (Experimental)
  Interventions: Other: Spencer technique along with conventional treatment
- Gongs Mobilization along with conventional treatment (Experimental)
  Interventions: Other: Gongs Mobilization along with conventional treatment

INTERVENTIONS:
Other: Spencer technique along with conventional treatment — Subjects in this group will receive conventional exercises and 7 stages of Spencer technique: (A) extension, (B) flexion, (C) circumduction with compression, (D) circumduction with traction, (E) abduction, (F) internal rotation, (G) lymphatic pump.
  Spencer technique will be used to increase range of motion of the glenohumeral joint. The patient will be positioned lying on the side with the affected shoulder above. The therapist will stabilize the shoulder girdle with the proximal hand and the distal hand will provide force into the restrictive barrier of shoulder in 7 different movements. These will be shoulder extension, circumduction with distraction, abduction, adduction with internal rotation and glenohumeral pump. During all the movements, patient will be asked to use muscle energy against the slight resistance offered by the therapist for 3-5 seconds. The exercise will be repeated 3-5 times with rest intervals over 3 sessions per week on alternate days for 4 weeks.
  Arms: Spencer technique along with conventional treatment
Other: Gongs Mobilization along with conventional treatment — The Gong's mobilization can be done either in high sitting or in side-lying position with the affected shoulder upward. The subject's shoulder will be abducted at 90° so that the humerus will be maintained at vertical position. The elbow joint will be flexed and maintained at 90°; the therapist will maintain this position by placing his/her hand below the subject's elbow. The humeral head will be pressed from anterior to posterior direction with the other hand. The therapist will hold the vertical axis of the humerus by maintaining the shoulder in abduction and the elbow in 90°. The therapist will raise his own body by slightly pulling on the anterior capsule and this pull will be maintained for 10-15 seconds and then relax for five seconds and will be performed for about two to three minutes. At this moment the subject will be asked to perform shoulder abduction with no external rotation, while elbow flexion will be maintained throughout.
  Arms: Gongs Mobilization along with conventional treatment

SUMMARY:
Adhesive capsulitis can be defined as insidious and progressive loss of both active and passive shoulder mobility in the glenohumeral joint presumably due to capsular contracture. It is associated with inflammation and stiffness of the capsule surrounding the glenohumeral joint, greatly restricting motion and causing chronic pain. The objective of this study is to compare the effects of spencer technique and gongs mobilization on pain, range of motion, disability, and scapular symmetry in patients with phase II adhesive capsulitis.

This study will be a Randomized Clinical trial involving 48 patients both males and females aged 40 to 60 years clinically diagnosed cases of phase II adhesive capsulitis. Patients will be randomly assigned into two groups using consecutive sampling technique. Group A will be treated with conventional treatment and spencer technique whereas Group B will be treated with conventional treatment and gongs mobilization. Numeric Pain Rating Scale will be used to measure pain of patients. Shoulder Pain and Disability Index score will be used to ask some questions related to patient's symptoms and disability. Lateral scapular slide test will be used to measure scapular symmetry and universal goniometer will be used to measure range of motion of shoulder joint. Each session will be repeated for 40 minutes thrice a week. All participants of the study will fill the Numeric Pain Rating Scale and Shoulder Pain and Disability Index score on day 1 as pretreatment values and at the end of 4th week as post treatment values respectively. The collected data will be analyzed on SPSS - 25.

Key words: Adhesive, scapula, mobilizations, glenohumeral joint, pain

DETAILED DESCRIPTION:
Adhesive capsulitis is characterized by a painful, gradual loss of both active and passive glenohumeral motion resulting from progressive fibrosis and ultimate contracture of the glenohumeral joint capsule. The term "frozen shoulder" was first introduced by Codman in 1934. He described frozen shoulder as a painful shoulder condition of insidious onset that was associated with stiffness and difficulty in sleeping on the affected side. In the general population, the incidence of adhesive capsulitis is 2-5%, more in females, those aged 40-65 years and those suffering from diabetes mellitus. In Pakistan, its precise prevalence is unknown, but, in general, it ranges 2-5%.

An increased incidence of frozen shoulder has been noticed in patients with hyperthyroidism and hypertriglyceridemia. Frozen shoulder progressive through three clinical phases painful phase- severe pain usually worst at night and when lying on the affected side (2-9 months) are stiffening or frozen phase- difficulty with simple activities of daily living. Stiffness progresses and leads to disused atrophy (4-12 months) Thawing phase - gradual increase in range of motion and improvement in pain, although it may reappear as stiffness ceases (5-12 months). In pathological condition like adhesive capsulitis where there is presence of capsular pattern of glenohumeral joint, in such a condition it is not possible to achieve full abduction through elevation because of marked limitation of external rotation.

Adhesive capsulitis is primarily categorized into two types: primary and secondary. Primary or idiopathic adhesive capsulitis is characterized by a gradual onset of pain and stiffness at the gleno-humeral joint without a specific cause. Secondary adhesive capsulitis is known to be caused by several predisposing factors. Women are affected more than men with a ratio of 58:423. The spencer technique is developed by spencer D. O. in 1916. This approach is a well-known osteopathic manipulative technique that focuses on mobilization of the glenohumeral and scapulothoracic joints. It helps the restricted joints to improve their functions, as well as positively affects other emotional, social, and cognitive areas. Spencer technique is an articulatory technique with 6 different procedures used to treat shoulder restriction caused by adhesive capsulitis. In this technique passive, smooth, rhythmic motion is designed to stretch contracted muscles, ligaments and capsules.

Physiotherapy methods such as active and active assisted exercises, pendular exercises, wand exercises, wall and ladder exercises, capsular stretching exercises and shoulder joint mobilization are often standard exercises in treating frozen shoulder. Electrotherapy modalities such as application of ultrasound, short-wave diathermy and LASER are used to relieve pain and promote hyperthermic effect to tissues.

Joint Mobilization is a manual therapy that applies passive traction and gliding motion to the articular surface to maintain free mobility of joints or to restore the normal condition of joints . Gong's mobilization technique helps to heal physical pain as well as distract the mind from stress. It is a corrective antero-posterior glide applied for shoulder distraction and their restricted movements to decrease pain and to improve range of motion. According to Wontae gong, gong's mobilization is more effective for anterior to posterior glide to improve shoulder abduction, external and internal rotation. Joint mobilization technique is effective to reduce pain and improves range of motion.

Many treatments have been advocated for Adhesive capsulitis: rest, analgesia, active and passive mobilization, physical therapy, oral and injected corticosteroids, capsular distension, manipulation under anesthesia, and arthroscopic capsular release. Currently, there is no consensus as to which is the most effective treatment. Evidence is present to support the isolated use of spencer technique on pain in adhesive capsulitis and isolated effects of gongs mobilizations on pain and disability in phase II adhesive capsulitis, while this study will determine the additional clinical evidence regarding the comparison of spencer technique and gongs mobilization on pain, range of motion, disability, and scapular symmetry in patients with phase II adhesive capsulitis to provide a better treatment option.

Adhesive Capsulitis is a commonest musculoskeletal problem affecting middle-aged person characterized by shoulder pain that is aggravated by movements and limitation of range of shoulder motion and daily activities. Adhesive capsulitis, is an idiopathic disease characterized by fibrosis, decreased volume of the glenoid capsule, and progressive pain with loss of range of motion (ROM). Shoulder pain and stiffness are accompanied by severe disability.

Rajalaxmi.V, S. Vasanthi, S.Sathya conducted a study in 2021 on the efficacy of Dynamic exercise and closed kinematic exercise combined with stretching in adhesive capsulitis. In this study concluded that s both the groups showed improvement while the Group (dynamic exercise with stretching) is more effective in reducing pain and disability than the Group (closed kinematic exercise with stretching) in adhesive capsulitis.

Mushyyaida Iqbal and colleagues in 2020 conducted a study to compare the effects of Spencer muscle energy technique and passive stretching in adhesive capsulitis. Spencer's joint mobility and muscle energy technique was found to be more effective than passive stretching exercises to reduce pain, and to improve joint ROM and functionality in AC.

Samiksha Sathe, Sukhna Kaur Khurana and coworkers conducted a study in 2018. The aim of that study was to compare the effect of Maitland mobilization as an intervention to conventional physiotherapy in patients with adhesive capsulitis on pain, ROM (flexion, abduction, external rotation, internal rotation) and Shoulder pain, and Disability Index (SPADI). On the basis of this study, it can be concluded that there is a more significant increase in ROM, and SPADI score, and a significant decrease in pain on NPRS by Maitland mobilization therapy along with conventional therapy as compared to conventional physiotherapy alone.

In 2017, a comparative study was done by Manish K. Sah, *Nagaraj, S. and Pearlson, K. according to that study, Gong's mobilization and Cyriax manipulation is equally effective in improving shoulder abduction and decreasing the functional deficit in subjects with frozen shoulder. According to Wontae Gong, in Gong's mobilization, abduction of the shoulder joint occurs when the humeral head is in normal position and the normal muscular contraction occurs with the rolling and sliding occurring at the articular surface and the tension of posterior joint capsule is reduced. And Gong's mobilization also corrects glenohumeral malalignment that can induce proper acceleration during treatment .

A randomized clinical trial was done in 2015 by Héctor Joaquín Gutiérrez Espinoza on short-term efficacy of a glenohumeral posterior mobilization technique versus conventional physiotherapy for the improvement of the range of external rotation in patients with primary adhesive capsulitis of the shoulder. The glenohumeral posterior mobilization technique applied after training with cycle ergometer is an effective short-term technique to treat primary adhesive capsulitis decreasing the severity of pain and improving joint function compared with conventional physiotherapy treatment. The degree of increase in shoulder external rotation is more than 20 degrees beyond the increase achieved with conventional treatment.

The literature has proved that muscle energy techniques and shoulder joint mobilizations are effective in reducing pain and stiffness in frozen shoulder (adhesive capsulitis) associated with scapular asymmetry. But spencer technique and gongs mobilizations are not compared before in treatment of scapular asymmetry associated with phase II adhesive capsulitis. As pain due to stiff shoulder in adhesive capsulitis may lead towards scapular asymmetry. Hence this study aims to compare the effects of spencer technique and gongs mobilization on pain, range of motion, disability, and scapular symmetry in patients with phase II adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age group between 40-60 years.
2. Both Males and Females.
3. Clinically diagnosed patients of phase II adhesive capsulitis will be included.
4. Adhesive Capsulitis subjects with limited Range of motion of shoulder abduction and external rotation.
5. Subjects with bilateral/unilateral adhesive capsulitis.

Exclusion Criteria:

1. Recent history of surgery on particular shoulder.
2. Patients with rotator cuff tears.
3. Rheumatoid and gouty arthritis.
4. Tumors of the shoulder region.
5. Subjects with acute inflammation.
6. Recent shoulder dislocation

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE | 4 weeks
  Numeric pain rating scale is a measurement of pain intensity in adults. The NPRS is a segmented numeric version of visual analogue scale (VAS) in which respondent select a whole number (0 to 10) that best reflects the intensity of pain. Scores range from 0 to 10
SHOULDER PAIN AND DISABILITY INDEX (SPADI) | 4 weeks
  SPADI 5 is a self-administered, shoulder-specific, fixed object index composed of 13 items divided into two subscales: pain (five items) and impairment (eight items). Responses to each item were recorded on a 10 point Likert scale, where 0= no pain or no difficulty and 10 =worst imaginable pain or so difficult it required help for the pain and disability items, respectively. The SPADI score is calculated by summing and then averaging the items of the two subscales to give a score out of 100 (higher scores reflects more pain/disability). The SPADI has acceptable test-retest reliability (intraclass correlation coefficients of 0.91 and 0.65 (95% CI, 0.42 to 0.8) in surgical and primary care populations respectively) and acceptable responsiveness
LATERAL SCAPULAR SLIDE TEST | 4 weeks
  Three positions are measured with the LSST designed by Kibler, is used to assess the scapular asymmetry under varying loads. To maintain a consistent posture during the various test positions, participants are instructed to fix their eyes on an object in the examination area. First test position, the participant is instructed to keep the arms relaxed at his/her sides, the most inferior aspect of the inferior angle of the scapula and the closest spinous process in the same horizontal plane is identified through palpation and marked. The distance between the 2 reference points is measured bilaterally with the help of a tape measure. This procedure is repeated for test position 2 (participant actively placed both hands on the ipsilateral hips, and consequently the humerus is positioned in medial rotation at -45° of abduction in the coronal plane) and test position 3 (the participant is instructed to maintain thumbs down position
UNIVERSAL GONIOMETER | 4 weeks
  Active and passive abduction (in the frontal plane) and external rotation (with the arm at 0 degrees of abduction) ROM measured with a conventional goniometer as per the guidelines given by the American Academy of Orthopedic Surgeons. Goniometric measurements are highly reliable provided measurements are conducted by same therapist (test-retest reliability: 0.94-0.98)

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah Rehabilitation Center, Lahore, Punjab Province
  - DHQ Hospital, Sheikhupura, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iqbal M, Riaz H, Ghous M, Masood K. Comparison of Spencer muscle energy technique and Passive stretching in adhesive capsulitis: A single blind randomized control trial. J Pak Med Assoc. 2020 Dec;70(12(A)):2113-2118. doi: 10.5455/JPMA.23971. PMID 33475581
- [Background] Nakandala P, Nanayakkara I, Wadugodapitiya S, Gawarammana I. The efficacy of physiotherapy interventions in the treatment of adhesive capsulitis: A systematic review. J Back Musculoskelet Rehabil. 2021;34(2):195-205. doi: 10.3233/BMR-200186. PMID 33185587
- [Background] Gutierrez Espinoza HJ, Pavez F, Guajardo C, Acosta M. Glenohumeral posterior mobilization versus conventional physiotherapy for primary adhesive capsulitis: a randomized clinical trial. Medwave. 2015 Sep 22;15(8):e6267. doi: 10.5867/medwave.2015.08.6267. English, Spanish. PMID 26485477
- [Background] Agarwal S, Raza S, Moiz JA, Anwer S, Alghadir AH. Effects of two different mobilization techniques on pain, range of motion and functional disability in patients with adhesive capsulitis: a comparative study. J Phys Ther Sci. 2016 Dec;28(12):3342-3349. doi: 10.1589/jpts.28.3342. Epub 2016 Dec 27. PMID 28174448